CLINICAL TRIAL: NCT03365635
Title: "Real World" Administration of Zepatier (Grazoprevir Plus Elvasvir) in Chronic Hemodialysis Patients With Hepatitis C Infection. Strategies for Identification of Patients, Insurance Approval, Treatment , and Laboratory Monitoring
Brief Title: Administration of Zepatier (Grazoprevir Plus Elbasvir) in Chronic Hemodialysis (HD) Patients With Hepatitis C
Acronym: HD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Michael Rudnick, Principle Investigator, University of Pennsylvania
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 828322
Record Dates: First submitted 2017-11-29; First posted 2017-12-07 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Hepatitis C; Hemodialysis; Nosocomial Infection
MeSH Terms: conditions — Hepatitis C; Cross Infection | interventions — elbasvir; grazoprevir; elbasvir-grazoprevir drug combination; Ribavirin

STUDY DESIGN:
Intervention Model Description: An interventional, prospective, non-randomized, non-blinded trial to evaluate real world strategies to identify and treat hepatitis C infected hemodialysis patients with Zepatier
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Genotype 1a -Rx naive -no NS5A polymorph (Experimental): Genotype 1a - treatment naive without NS5A polymorphism - Drug Intervention : Oral administration Elbasvir (50mg)/Grazoprevir (100mg) one tablet per day for 12 weeks
  Interventions: Drug: Elbasvir 50 MG / Grazoprevir 100 MG [Zepatier]
- Genotype 1a, Rx naive + NS5A polymorph (Experimental): Genotype 1a - treatment naiive with NS5A polymorphism - Oral administration of Elbasvir/Grazoprevir one tablet daily and ribavirin (200 mg) daily for 16 weeks weeks
  Interventions: Drug: Elbasvir 50 MG / Grazoprevir 100 MG [Zepatier]
- Genotype 1b - Rx naive (Experimental): Genotype 1b-treatment naive - Oral administration of Elbasvir/Grazoprevir one daily for 12 weeks
  Interventions: Drug: Elbasvir 50 MG / Grazoprevir 100 MG [Zepatier]
- Genotype 1a/1b -prior INF or NS3/4A (Experimental): Genotype 1a or 1b - prior treatment with INF or HCV NS3/4A protease inhibitor - oral administration of Elbasvir/Grazoprevir and ribavirin each once daily for 12 weeks
  Interventions: Drug: Elbasvir 50 MG / Grazoprevir 100 MG [Zepatier]
- Genotype4 - treatment naive (Experimental): (e) Genotype 4 - treatment naive - oral administration of Elbasvir/Grazoprevir one daily for 12 weeks
  Interventions: Drug: Elbasvir 50 MG / Grazoprevir 100 MG [Zepatier]
- Genotype 4- prior treatment (Experimental): Genotype 4 -prior treatment - oral administration of Elbasvir/Grazoprevir and ribavirin each once per day for 16 weeks
  Interventions: Drug: Elbasvir 50 MG / Grazoprevir 100 MG [Zepatier]

INTERVENTIONS:
Drug: Elbasvir 50 MG / Grazoprevir 100 MG [Zepatier] — Same as described in arm description
  Other Names: Ribavirin 200 mg

SUMMARY:
This is a study to define strategies for Nephrologists to directly supervise and apply direct acting antivirals to cure hepatitis C in hemodialysis patients. Strategies will include identification of candidate patients, application for insurance approval, specifics of direct acting antiviral therapy (Zepatier with or without ribavirin) and laboratory monitoring during and after therapy.

DETAILED DESCRIPTION:
Background - Hepatitis C (HCV) is common in hemodialysis (HD) patients with reported prevalences of 25%, By 2020, predicted 775,000 hemodialysis patients in the US, of whom 109,000 will have HCV. Hepatitis C is associated with increased mortality in HD patients, decreased kidney allograft survival, and a source of nosocomial infection in hemodialysis units. Currently drugs to cure HCV - direct acting antivirals (DAA) which can be safely given to HD patients are now available. A significant portion of the medical care provided to HD patients is by Nephrologists and HD staff.

Goals of Protocol - 1. Provide guidelines for implementation and monitoring of DAA therapy in HD patients with HCV 2. Provide Nephrologists strategies for identification of candidate HD patients, obtainment of third party approval for DAA payment, specific drug dosing protocols based on genome type of HCV, and laboratory and clinical monitoring during DDA therapy. 3, By reducing the pool of HCV patients in a HD Unit, the risk of nosocomial transmission of HCV t o other patients and staff will be reduced

Study Design - an interventional, prospective, non-randomized, non-blinded trial to evaluate real world strategies to identify and treat HCV infected patients with Zepatier

Study Procedures 1. Patients who meet inclusion criteria without exclusion criteria be assigned treatment with Zepatier with or without Ribavirin according to following schedule: (a) Genotype 1a - treatment naive without NS5A polymorphism - Zepatier one tablet (100 mg grazoprevir and 50 mg elbasvir) per day for 12 weeks (b) Genotype 1a - treatment naiive with NS5A polymorphism - Zepatier one tablet daily and ribavirin (200 mg) daily for 16 weeks (c) Genotype 1b-treatment naive - Zepatier one daily for 12 weeks (d) Genotype 1a or 1b - prior treatment with INF or HCV NS3/4A protease inhibitor - Zepatier and ribavirin each once daily for 12 weeks (e) Genotype 4 - treatment naive - Zepatier one daily for 12 weeks (f)Genotype 4 -prior treatment - Zepatier and ribavirin each once per day for 16 weeks

Baseline/Screening Testing: 1. HCV genotype testing 2. HCV viral RNA load 3. Liver function tests 4, Protime, Partial Thromboplastin time 5. HIV - if positive, then determine viral RNA and CD4 and T cell count 6. Liver biopsy (within 24 mo of treatment) or Fibroscan within 12 mo of treatment 7. Hepatitis BsAg 8. For patients with HCV genotype 1a, test fro NS5A mutation

Treatment of HIV/HCV co-infected patients will be done in collaboration with the HIV treating physician to determine if any adjustments in the HIV drug regimen will be required

Testing/Evaluations during Active DAA Treatment - 1. LFT and RNA HCV viral load at week 4, 8, and 12. For patients on 16 weeks of treatment, LFT at week 16 as well 2. For patients on combination Zepatier and ribavirin, hemoglobin monitoring every week during treatment 3. Clinical pharmacology evaluation for compliance and adverse events at week 4,8,and 12 (and week 16 for patients on 16 week treatment)

Testing/Evaluation Post DAA Treament - 1, RNA viral load at 12 weeks post treatment 2. Clinical Pharmacologoy evaluation 12 weeks post treatment for adverse events 3. patients who achieve sustained viral remission at 12 weeks will be identified in HD records as HCV ab positive but HCV viral load RNA negative

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patient
* > age 18 years old
* Hepatitis C antibody positive and Hepatitis C RNA Quantification positive
* Hepatitis C genomes 1a, 1b, or 4
* Prior Interferon , ribavirin treatment failures , partial responders, or intolerance to these treatment allowed to enroll
* Not of reproductive potential - hemodialysis patients must have no menses for 12 months
* Males with partners of reproductive potential as along a 2 reliable forms of contraception are used simultaneously during treatment and for 6 months after completion of treatment
* Ability to understand the study procedures, alternative treatments available, risks of participating in the study, and voluntarily agree to participate

Exclusion Criteria:

* Currently undergoing active treatment for HCV with a direct acting antiviral or have previously successfully been treated with a direct acting antiviral
* Have moderate or severe hepatic disease - Child-Pugh B or C
* Have evidence of decompensated liver disease manifested by ascites, gastric or variceal bleeding, hepatic encephalopathy, or other signs/symptoms of advanced liver disease
* Co-administration of known heaptotoxic drugs including but not limited to : etofoxine, isoniazid, nitrofurantoin, phenytoin
* Use of strong CYP3A/P-gp inhibitors, organic acid transporting polypeptide 1B1/3 inhibitors, strong inducers of cytochrome 450 3A (CYP3A), efavirenz, or other drugs which may interact with elbasvir/grazoprevir as per package insert
* history of substance abuse with alcohol, intravenous drugs, psychotropics, narcotics, cocaine use within 1 year of screening for study
* history of any condition, pre-study lab abnormality, or ECG abnormality or history of any illness which in the opinion of the investigators might confound the results of the study or pose additional risks from the administration of elbasvir/grazoprevir
* Have evidence of history of chronic hepatitis not caused by HCV including but not limited to nonalcoholic steatohepatitis (NASH), drug induced hepatitis, and autoimmune hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-22 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Rudnick, MD, Principal Investigator — University of Pennsylvania Health System
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No research reason to share IPD to other researchers

REFERENCES:
- [Background] Roth D, Nelson DR, Bruchfeld A, Liapakis A, Silva M, Monsour H Jr, Martin P, Pol S, Londono MC, Hassanein T, Zamor PJ, Zuckerman E, Wan S, Jackson B, Nguyen BY, Robertson M, Barr E, Wahl J, Greaves W. Grazoprevir plus elbasvir in treatment-naive and treatment-experienced patients with hepatitis C virus genotype 1 infection and stage 4-5 chronic kidney disease (the C-SURFER study): a combination phase 3 study. Lancet. 2015 Oct 17;386(10003):1537-45. doi: 10.1016/S0140-6736(15)00349-9. Epub 2015 Oct 5. PMID 26456905
- [Background] Goodkin DA, Bieber B, Jadoul M, Martin P, Kanda E, Pisoni RL. Mortality, Hospitalization, and Quality of Life among Patients with Hepatitis C Infection on Hemodialysis. Clin J Am Soc Nephrol. 2017 Feb 7;12(2):287-297. doi: 10.2215/CJN.07940716. Epub 2016 Dec 1. PMID 27908905
- [Background] Zaki MSE. The effect of Hepatitis C Virus infection on cardiovascular complications in end stage kidney disease patients on regular hemodialysis. Electron Physician. 2017 Feb 25;9(2):3857-3861. doi: 10.19082/3857. eCollection 2017 Feb. PMID 28465818
- [Background] Jadoul M, Horsmans Y. Towards eradication of hepatitis C virus from dialysis units. Lancet. 2015 Oct 17;386(10003):1514-5. doi: 10.1016/S0140-6736(15)00381-5. Epub 2015 Oct 5. No abstract available. PMID 26456906
- [Background] Lo Re V. Extrahepatic Complications of Hepatitis C Virus Infection in HIV and the Impact of Successful Antiviral Treatment. Clin Infect Dis. 2017 Feb 15;64(4):498-500. doi: 10.1093/cid/ciw814. No abstract available. PMID 28172488
- [Background] Cacoub P, Desbois AC, Isnard-Bagnis C, Rocatello D, Ferri C. Hepatitis C virus infection and chronic kidney disease: Time for reappraisal. J Hepatol. 2016 Oct;65(1 Suppl):S82-S94. doi: 10.1016/j.jhep.2016.06.011. PMID 27641990
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO). KDIGO clinical practice guidelines for the prevention, diagnosis, evaluation, and treatment of hepatitis C in chronic kidney disease. Kidney Int Suppl. 2008 Apr;(109):S1-99. doi: 10.1038/ki.2008.81. No abstract available. PMID 18382440
- [Background] Rao AK, Luckman E, Wise ME, MacCannell T, Blythe D, Lin Y, Xia G, Drobeniuc J, Noble-Wang J, Arduino MJ, Thompson ND, Patel PR, Wilson LE. Outbreak of hepatitis C virus infections at an outpatient hemodialysis facility: the importance of infection control competencies. Nephrol Nurs J. 2013 Mar-Apr;40(2):101-10, 164; quiz 111. PMID 23785746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients from an outpatient hemodialysis unit were recruited between October 2019 and April 2020
Pre-assignment Details: There was no wash out or run-in period to this protocol
Period: Overall Study
Arm/Group | Genotype 1a -Rx Naive -no NS5A Polymorph | Genotype 1a, Rx Naive + NS5A Polymorph | Genotype 1b - Rx Naive | Genotype 1a/1b -Prior INF or NS3/4A | Genotype4 - Treatment Naive | Genotype 4- Prior Treatment
Started | 3 | 0 | 1 | 0 | 0 | 0
Completed | 3 | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Genotype 1a, Rx naive + NS5A polymorph, Genotype 1a/1b - prior INF or NS3/4A, Genotype 4- treatment naive and prior treatment - none of the recruited patients fell into these categories after initial screening
Groups:
- Total: Total of all reporting groups
Arm/Group | Genotype 1a -Rx Naive -no NS5A Polymorph | Genotype 1a, Rx Naive + NS5A Polymorph | Genotype 1b - Rx Naive | Genotype 1a/1b -Prior INF or NS3/4A | Genotype4 - Treatment Naive | Genotype 4- Prior Treatment | Total
Number analyzed (Participants) | 3 | 0 | 1 | 0 | 0 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 |  | 0 | 0 | 0 | 0 | 0
  >=65 years | 3 | 0 | 1 | 0 | 0 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 0 |  |  |  | 1
  Male | 2 |  | 1 |  |  |  | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 |  |  |  | 0
  Asian | 0 |  | 0 |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 |  |  |  | 0
  Black or African American | 3 |  | 1 |  |  |  | 4
  White | 0 |  | 0 |  |  |  | 0
  More than one race | 0 |  | 0 |  |  |  | 0
  Unknown or Not Reported | 0 |  | 0 |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 1 |  |  |  | 4

OUTCOME MEASURES:

1. Primary Outcome: SVR - Sustained Virologic Response
Description: Absence of HCV by viral RNA quantitation at 12 weeks post treatment
Time Frame: 12 weeks after completion of Elbasivir/Grazoprevir treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype 1a -Rx Naive -no NS5A Polymorph | Genotype 1a, Rx Naive + NS5A Polymorph | Genotype 1b - Rx Naive | Genotype 1a/1b -Prior INF or NS3/4A | Genotype4 - Treatment Naive | Genotype 4- Prior Treatment
Number analyzed (Participants) | 3 | 0 | 1 | 0 | 0 | 0
Participants | 3 | 0 | 1 | 0 | 0 |

2. Secondary Outcome: Approval for DAA by Third Party Payers
Description: The number of participants for whom their third party insurance approved payment of the DAA (study drug)
Time Frame: Within one month of last patient enrolled
Population: No patients were recruited into some of the subgroups and this is noted as 0 participants for these subgroups
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype 1a -Rx Naive -no NS5A Polymorph | Genotype 1a, Rx Naive + NS5A Polymorph | Genotype 1b - Rx Naive | Genotype 1a/1b -Prior INF or NS3/4A | Genotype4 - Treatment Naive | Genotype 4- Prior Treatment
Number analyzed (Participants) | 3 | 0 | 1 | 0 | 0 | 0
Participants | 0 |  | 0 |  |  |

ADVERSE EVENTS:
Time Frame: 24 weeks from start of therapy
Description: No definitions different than clinicaltrials.gov definitions. No adverse events
Arm/Group | Genotype 1a -Rx Naive -no NS5A Polymorph | Genotype 1a, Rx Naive + NS5A Polymorph | Genotype 1b - Rx Naive | Genotype 1a/1b -Prior INF or NS3/4A | Genotype4 - Treatment Naive | Genotype 4- Prior Treatment
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0 | 0/1 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/1 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/1 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We anticipated screening 30 patients and enrolling 25 patients. However, there was a significant delay in the regulatory approvals for the protocol and during this delay period, many of the potential patients ultimately received direct acting antivirals from the primary care physicians or other physicians outside of Nephrology

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT03365635/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT03365635/SAP_001.pdf
  • Informed Consent Form (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT03365635/ICF_002.pdf